CLINICAL TRIAL: NCT06420635
Title: Effect of an Interdisciplinary Intervention Program on Maternal Self-efficacy and Motor Development of Premature Children: Clinical Trial Protocol
Brief Title: Maternal Self-efficacy and Motor Development in Premature Infants: Clinical Trial Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de la Sabana (Other)
Collaborators: Universidad de Boyacá (Other); Hospital Universitario de La Samaritana (Unknown); Universidade Franciscana (UFN)- Brasil (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENF-64-2022
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Premature Birth; Mothers of Newborn Infants
Keywords: Premature newborn; Mothers; self-efficacy; motor skills; motor praxis; outpatient care; information and communication technologies; kangaroo mother care; nursing; physical therapy
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interdisciplinary intervention program on maternal self-efficacy and motor development (Experimental): Interdisciplinary intervention program on maternal self-efficacy and the motor development of premature children.
  Interventions: Behavioral: Interdisciplinary intervention program on maternal self-efficacy and the motor development of premature children
- Traditional Kangaroo Program (Active Comparator): The control group will receive the conventional family-centered care plan, including kangaroo position, exclusive breastfeeding, and monitoring of the child's progress.
  Interventions: Behavioral: Traditional kangaroo program

INTERVENTIONS:
Behavioral: Interdisciplinary intervention program on maternal self-efficacy and the motor development of premature children — The experimental group will receive an intervention about maternal self-efficacy and motor stimulation strategies for premature children applied by mothers. There will be two face-to-face meetings: the first with a theoretical session on motor development, a practical workshop on stimulation skills using a baby simulator and strengthening of maternal self-efficacy. The second meeting seeks for mothers to reflect on self-efficacy and carry out practical simulation of strategies with their children. At home (for four weeks), self-efficacy will be strengthened through 4 strategies twice a week, for 8 sessions. Mothers will put into practice with the baby the 10 stimulation strategies explained in the face-to-face sessions, must complete 14 sessions per week, 2 times a day, for a total of 56 sessions. The initial measurement will be carried out before the intervention, the second at 4 weeks and the third at 8 weeks after the intervention began.
  Arms: Interdisciplinary intervention program on maternal self-efficacy and motor development
Behavioral: Traditional kangaroo program — The control group will receive the conventional family-centered care plan, including kangaroo position, exclusive breastfeeding, and outpatient follow-up. The traditional intervention for the control group is based on the Kangaroo Mother Method (KMC) program, proposed according to technical guidelines, which promotes skin-to-skin contact between mother and premature baby. In periodic outpatient consultations, clinical assessments are carried out focused on optimal growth (goal 15-20g/kg/day), neurological and psychomotor development, and timely detection of pathologies that require specialized care according to findings. Compliance with the vaccination schedule and medical indications, and assurance of breastfeeding, are monitored. The frequency of check-ups is daily initially, then weekly until 40 weeks and then monthly. The approach includes early stimulation and follow-up until 12 months of corrected age.
  Arms: Traditional Kangaroo Program

SUMMARY:
Mothers of premature newborns face special home care situations due to the conditions of their children after hospital discharge; This requires promoting the positive perception of maternal self-efficacy and thus achieving the reinforcement of behaviors related to the demand for care in relation to motor development.

* Objective: Determine the effect of an interdisciplinary intervention program on maternal self-efficacy and motor development of premature children in the cities of Bogotá and Tunja in comparison with the traditional kangaroo program.
* Methodology: Experimental study, with pretest/posttest design, with experimental and control group, which determines the baseline. With initial evaluation of the groups, randomized assignment, and post-intervention evaluation at 4 weeks and flow-up at 8 weeks. The intervention will be developed in two scenarios, in the outpatient kangaroo plan consultation and at home. The experimental group will receive an intervention based on the promotion of maternal self-efficacy and the motor development of the premature baby. The control group will have traditional kangaroo program care. The sample calculation is 92 participants, 46 in the experimental group and 46 in the control group. The intervention, evaluations and data analysis will be developed by blinded professionals. An analysis of the data will be done by intention to treat.
* Type of results expected to be obtained: It is expected to obtain an intervention that promotes maternal self-efficacy for the adequate stimulation of the motor development of the premature baby. It is expected to enhance the confidence and empowerment of the maternal role, the motor development of children in accordance with the corrected age and the incorporation of ICT for monitoring at home.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of a child born prematurely who attend the outpatient kangaroo mother program in Bogotá, Tunja and Zipaquirá in the period between 2024 and 2025.
* Premature children between 32 to 36.6 weeks who participate in the outpatient kangaroo mother program in Bogotá, Tunja and Zipaquirá in the period between 2024 and 2025.

Exclusion Criteria:

* Mothers who manifest any diagnosed mental limitation to participate in the study.
* Premature children with hemodynamic alterations, congenital malformations, chromosomal syndromes, esophageal atresia, ductus arteriovenosus, heart disease and neurological pathologies.

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Estimated)
Dates: Start 2024-06-25 (Estimated); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Maternal self-efficacy | Two months
  Parental Evaluation Scale (PES). The total score is 10, the minimum value is 0, and the maximum is 10. Higher scores indicate a greater perception of self-efficacy and maternal satisfaction.
Motor Development | Two months
  Alberta Infant Motor Scale (EMIA). The total score is 90, the minimum value is 5, and the maximum is 90. Higher scores indicate a greater motor development, which is directly proportional to the corrected age of children.

CONTACTS AND LOCATIONS:
Overall Officials: Angélica Ospina, PhD, Principal Investigator — Universidad de la Sabana

IPD SHARING:
Plan to Share IPD: No